CLINICAL TRIAL: NCT01527201
Title: Design of a Randomized Controlled Trial Examining the Effects of Arthroscopic Debridement on Chondral Lesions in Patients Undergoing Partial Meniscectomy: The ChAMP (Chondral Lesions And Meniscus Procedures) Trial
Brief Title: The ChAMP (Chondral Lesions And Meniscus Procedures) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leslie Bisson, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPS1561011B
Record Dates: First submitted 2012-01-19; First posted 2012-02-06 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Meniscal Tear; Chondromalacia
Keywords: Arthroscopy; Debridement
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): Worn out cartilage will be surgically treated.
  Interventions: Procedure: Arthroscopic debridement
- Control Group (No Intervention): Worn out cartilage will be observed, but will not be treated surgically.

INTERVENTIONS:
Procedure: Arthroscopic debridement — Surgeon will debride, or remove, worn out cartilage.
  Other Names: Chondroplasty
  Arms: Treatment Group

SUMMARY:
The purpose of this randomized controlled trial is to determine the effectiveness of treating cartilage lesions found during knee arthroscopy.

DETAILED DESCRIPTION:
Normal wear-and-tear on the knee can cause tissue, or cartilage, in the knee to soften over time forming chondral lesions. Worn out cartilage is often found during knee surgery for other conditions. Typically, surgeons will remove any worn out cartilage that is found using a procedure called debridement. However, the investigators do not know if surgically treating the worn out cartilage is better than leaving the tissue untreated, so it is necessary to compare the two. Patients who are found to have worn out cartilage during arthroscopy, will be randomly assigned to either receive treatment (debridement) or non-treatment (observation) of their cartilage. Patients without worn out cartilage will also be included in this study and observed postoperatively.

The primary objective of this study is to examine the effects of treatment of worn out cartilage (versus non-treatment of worn out cartilage and versus patients without worn out cartilage), on self-reported knee pain following arthroscopic meniscectomy using a double-blinded randomized controlled trial design. Secondary objectives of this study include examining the effects of treating worn out cartilage on other outcomes (subjective knee and general health scores and knee measurements including range of motion, presence of effusion and quadriceps circumference) and also to calculate the intra-operative costs associated with treatment, including the amount of time and instruments needed for debridement.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo a meniscectomy
* Patients with chondral lesions found during meniscectomy
* Patients without chondral lesions are not eligible for randomization to one of the study arms, but will still be included in the study and observed after surgery

Exclusion Criteria:

* Osteochondritis dissecans
* Large chondral flaps judged to be impending loose bodies
* Joint space loss of affected compartment greater than 50% compared to opposite side
* Visible osteophytes of the medial or lateral compartment
* Previous knee surgery on the affected side
* Previous major knee trauma
* History of inflammatory joint disease, gout, or chondrocalcinosis
* Presence of worker's compensation claim
* Patients undergoing meniscal repair
* Patients undergoing microfracture for contained grade IV chondral lesions
* Presence of significant ligamentous instability in the operative knee (i.e., complete acruciate ligament (ACL) or posterior cruciate ligament (PCL) tear, grade III medial or lateral side instability)
* Major neurologic deficit
* Serious medical illness with limited life expectancy or that poses high intraoperative risk
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2012-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Self-reported knee pain | 1-year after surgery

SECONDARY OUTCOMES:
Intra-operative costs associated with debridement (i.e., time and instruments needed to debride) | Measured during surgery
  Surgeon records and documents the time and instruments needed for debridement.
Subjective measures and knee measurements | 1-year after surgery
  Subjective knee and general health scores will be assessed. Also, knee measurements including range of motion, presence of effusion, and quadriceps circumference will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Bisson, MD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- UB Orthopaedics and Sports Medicine, Buffalo, New York, United States

REFERENCES:
- [Background] Kirkley A, Birmingham TB, Litchfield RB, Giffin JR, Willits KR, Wong CJ, Feagan BG, Donner A, Griffin SH, D'Ascanio LM, Pope JE, Fowler PJ. A randomized trial of arthroscopic surgery for osteoarthritis of the knee. N Engl J Med. 2008 Sep 11;359(11):1097-107. doi: 10.1056/NEJMoa0708333. PMID 18784099
- [Background] Moseley JB, O'Malley K, Petersen NJ, Menke TJ, Brody BA, Kuykendall DH, Hollingsworth JC, Ashton CM, Wray NP. A controlled trial of arthroscopic surgery for osteoarthritis of the knee. N Engl J Med. 2002 Jul 11;347(2):81-8. doi: 10.1056/NEJMoa013259. PMID 12110735